CLINICAL TRIAL: NCT05338866
Title: Chemotherapy Combined With High-dose Radiotherapy for Low Rectal Cancer Using Magnetic Resonance Guided Radiotherapy Linear Accelerator：A Prospective Phase 2 Trial
Brief Title: Chemotherapy Combined With High-dose Radiotherapy for Low Rectal Cancer Using MR Guided Linear Accelerator
Status: Enrolling by invitation | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Professor, Sun Yat-sen University
Other Study IDs: 2021-FXY-489
Record Dates: First submitted 2022-04-05; First posted 2022-04-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
Keywords: Lower rectal cancer; Magnetic resonance imaging guided radiation therapy; High-dose radiotherapy; Toxic and side effects; Quality of life score
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1. Cohort 2: A total of 6 courses of oxaliplatin plus capecitabine chemotherapy and 2 courses of capecitabine single drug chemotherapy were performed. Concurrent chemoradiotherapy starts at the second cycle.
  Cohort 1: For patients with low rectal cancer who refused surgery before the initial diagnosis and treatment, the first stage of radiotherapy used conventional linear accelerated radiotherapy, with doses of GTV 50Gy/25f and CTV 45Gy/25f for 5-6 weeks. Subsequently, the second stage of radiotherapy boost was continued with MR linear accelerator, and the dose was GTV 16~20Gy/8~10f for 2 weeks.
  Cohort 2: For locally advanced low rectal cancer patients who did not achieve clinical complete remission 6-8 weeks after neoadjuvant radiochemotherapy and refused surgery, radiotherapy was given in the first stage at the doses of GTV 50Gy/25f and CTV 45Gy/25f for 5-6 weeks. In the second stage, MR linear accelerator was used for radiotherapy boosting, and the dose was GTV 30Gy/15f for 3 weeks.
  Interventions: Radiation: Magnetic resonance guided radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Magnetic resonance guided radiotherapy — Radical radiotherapy boosting for low rectal cancer through magnetic resonance guided radiotherapy linear accelerator.
Drug: Chemotherapy — For patients with AJCC stage II and III and age < 72 years old, Capox ×6→capecitabine×2.
  Detailed usage: Oxaliplatin 130mg/m2 (reduced to 100mg/m2 during concurrent chemoradiotherapy), intravenous administration, d1. Capecitabine 1000mg / m2, twice a day, d1-14. Repeated every 3 weeks.
  For patients aged ≥ 72 years, or the competent physician judges that the patients cannot tolerate dual drug combined chemotherapy, capecitabine ×8 courses.
  For patients with AJCC stage I, capecitabine ×4 courses.
  Other Names: Capox, Capecitabine

SUMMARY:
The incidence rate of colorectal cancer is third in male tumors and second in female tumors. The newly diagnosed incidence of colorectal cancer is no less than 100 thousand in China, which poses a great threat to people's health and a heavy burden of public health. Preoperative neoadjuvant radiotherapy and chemotherapy combined with radical surgery is recommended for locally advanced rectal cancer. Low rectal cancer accounts for about one third of all rectal cancer cases. Due to the particularity of its location，surgical complications and postoperative patients need permanent colostomy (artificial anus) to solve the defecation problems, which has a serious impact on the patients' work and life. How to improve the quality of life of patients without reducing the survival rate has become an important topic in the treatment of low rectal cancer. Previous studies have shown that the prognosis of patients with pathological complete remission (pCR) after neoadjuvant chemoradiotherapy for rectal cancer is optimistic. The clinical efficacy of "observation and waiting" is good. The results of small sample exploratory clinical studies of radical radiotherapy and chemotherapy for low rectal cancer are satisfactory, and MR-linear accelerator can be used for precision radiotherapy for colorectal cancer.

This study is aimed to explore the efficacy and safety of radical radiotherapy boost for low rectal cancer by using magnetic resonance guided radiotherapy system, and further evaluate the impact of boost on the quality of life of patients.

DETAILED DESCRIPTION:
It is a prospective phase II, non-randomized controlled designed clinical study. For the optimal design, 58 cases of low rectal adenocarcinoma without metastasis were divided into queue 1 and queue 2 according to the start time of boost. MR-linear accelerator was used for dose boost of the local tumor region to make it reaching the radical radiotherapy dose. At the same time, fluorouracil based chemotherapy was given according to stages.

The primary endpoint was 3-year progression free survival rate. The secondary end points were 3-year stoma free survival rate, 3-year local regeneration rate, 3-year disease-free survival rate, 3-year distant metastasis rate, 3-year overall survival rate, short term and long-term toxic and side effects, and patients' quality of life scale 1-3 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed as rectal adenocarcinoma.
2. MRI and / or electronic colonoscopy confirmed that the lower edge of the tumor was ≤ 5cm from the anal edge.
3. The AJCC clinical stage was cT1-4NxM0, with or without MRF positive and EMVI positive.
4. MSI gene detection or MMR protein immunohistochemical detection was MSS / PMMR.
5. No obvious signs of intestinal obstruction or intestinal obstruction has been relieved after proximal colostomy.
6. Age: 18 ~ 80 years old.
7. ECOG score: 0-1.
8. Expected life: more than 3 years.
9. Hematology: WBC > 3 × 109/L; PLT>80 × 109/L; Hb>90g/L.
10. Liver function: ALT and AST were less than 2 times of normal value; Bilirubin is less than 1.5 times of normal value.
11. Renal function: creatinine is less than 1.5 times of normal value or creatinine clearance rate (CCR) ≥ 60ml / min.
12. Patient who has not received tumor resection, radiotherapy, chemotherapy, immunotherapy or other anti-tumor treatment.

Exclusion Criteria:

1. There are any conditions that make MRI impossible.
2. There are serious medical complications.
3. Uncontrolled infectious diseases, autoimmune diseases and mental diseases.
4. Any unstable condition or situation that may endanger patient safety and compliance.
5. Pregnant or lactating women who are fertile and do not take adequate contraceptive measures.
6. Refuse to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower rectal cancer who refuse surgery for various reasons or are not suitable for surgery due to systemic diseases.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year progression free survival rate | 3-year after enrollment
  Percentage of survive patients with no disease progression or death after 3 years from enrollment.

SECONDARY OUTCOMES:
3-year stoma free survival rate | 3-year after enrollment
  Percentage of patients survive with no enterostomy after 3 years from enrollment.
3-year local regeneration rate | 3-year after enrollment
  Percentage of patients with no local tumor regeneration after 3 years from enrollment.
3-year disease-free survival rate | 3-year after enrollment
  The percentage of patients survive with no disease after 3 years from enrollment
3-year distant metastasis rate | 3-year after enrollment
  The percentage of patients with distant metastasis.
3-year overall survival rate | 3-year after enrollment
  The percentage of patients survive 3 years after enrollment
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | During treatment. 3-month, 6-month, 1-year, 3-year after treatment.
  Acute and chronic toxic and side effects
Patients' quality of life scale | Before and during treatment. 3-month, 6-month, 1-year, 3-year after enrollment.
  Patients' quality of life scale

CONTACTS AND LOCATIONS:
Overall Officials: Yuanhong Gao, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Study data can be shared after publication of the study results, upon request.

REFERENCES:
- [Background] Wang Q, Zhang S, Zhou C, et al. Efficacy and safety of high dose radiotherapy for the treatment of locally advanced rectal cancer. International Journal of Radiation Oncology Biology Physics. 2020. 108(3): e644-e645
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Result] Glimelius B, Tiret E, Cervantes A, Arnold D; ESMO Guidelines Working Group. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi81-8. doi: 10.1093/annonc/mdt240. No abstract available. PMID 24078665
- [Result] Galandiuk S, Wieand HS, Moertel CG, Cha SS, Fitzgibbons RJ Jr, Pemberton JH, Wolff BG. Patterns of recurrence after curative resection of carcinoma of the colon and rectum. Surg Gynecol Obstet. 1992 Jan;174(1):27-32. PMID 1729745
- [Result] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Result] Heald RJ, Ryall R. Recurrent cancer after restorative resection of the rectum. Br Med J (Clin Res Ed). 1982 Mar 13;284(6318):826-7. doi: 10.1136/bmj.284.6318.826-e. No abstract available. PMID 6802248
- [Result] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Result] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Result] Roh MS, Colangelo LH, O'Connell MJ, Yothers G, Deutsch M, Allegra CJ, Kahlenberg MS, Baez-Diaz L, Ursiny CS, Petrelli NJ, Wolmark N. Preoperative multimodality therapy improves disease-free survival in patients with carcinoma of the rectum: NSABP R-03. J Clin Oncol. 2009 Nov 1;27(31):5124-30. doi: 10.1200/JCO.2009.22.0467. Epub 2009 Sep 21. PMID 19770376
- [Result] Benson AB 3rd, Venook AP, Bekaii-Saab T, Chan E, Chen YJ, Cooper HS, Engstrom PF, Enzinger PC, Fenton MJ, Fuchs CS, Grem JL, Grothey A, Hochster HS, Hunt S, Kamel A, Kirilcuk N, Leong LA, Lin E, Messersmith WA, Mulcahy MF, Murphy JD, Nurkin S, Rohren E, Ryan DP, Saltz L, Sharma S, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Gregory KM, Freedman-Cass D. Rectal Cancer, Version 2.2015. J Natl Compr Canc Netw. 2015 Jun;13(6):719-28; quiz 728. doi: 10.6004/jnccn.2015.0087. PMID 26085388
- [Result] Sautter-Bihl ML, Hohenberger W, Fietkau R, Rodel C, Schmidberger H, Sauer R. Rectal cancer : when is the local recurrence risk low enough to refrain from the aim to prevent it? Strahlenther Onkol. 2013 Feb;189(2):105-10. doi: 10.1007/s00066-012-0299-5. PMID 23299826
- [Result] Feddern ML, Emmertsen KJ, Laurberg S. Life with a stoma after curative resection for rectal cancer: a population-based cross-sectional study. Colorectal Dis. 2015 Nov;17(11):1011-7. doi: 10.1111/codi.13041. PMID 26112651
- [Result] Konanz J, Herrle F, Weiss C, Post S, Kienle P. Quality of life of patients after low anterior, intersphincteric, and abdominoperineal resection for rectal cancer--a matched-pair analysis. Int J Colorectal Dis. 2013 May;28(5):679-88. doi: 10.1007/s00384-013-1683-z. Epub 2013 Apr 10. PMID 23571868
- [Result] Lim L, Chao M, Shapiro J, Millar JL, Kipp D, Rezo A, Fong A, Jones IT, McLaughlin S, Gibbs P. Long-term outcomes of patients with localized rectal cancer treated with chemoradiation or radiotherapy alone because of medical inoperability or patient refusal. Dis Colon Rectum. 2007 Dec;50(12):2032-9. doi: 10.1007/s10350-007-9062-x. Epub 2007 Sep 26. PMID 17896138
- [Result] Gao YH, Lin JZ, An X, Luo JL, Cai MY, Cai PQ, Kong LH, Liu GC, Tang JH, Chen G, Pan ZZ, Ding PR. Neoadjuvant sandwich treatment with oxaliplatin and capecitabine administered prior to, concurrently with, and following radiation therapy in locally advanced rectal cancer: a prospective phase 2 trial. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):1153-60. doi: 10.1016/j.ijrobp.2014.07.021. Epub 2014 Oct 13. PMID 25442042
- [Result] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Result] Habr-Gama A, Perez RO, Nadalin W, Sabbaga J, Ribeiro U Jr, Silva e Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Operative versus nonoperative treatment for stage 0 distal rectal cancer following chemoradiation therapy: long-term results. Ann Surg. 2004 Oct;240(4):711-7; discussion 717-8. doi: 10.1097/01.sla.0000141194.27992.32. PMID 15383798
- [Result] Habr-Gama A, Perez RO, Proscurshim I, Campos FG, Nadalin W, Kiss D, Gama-Rodrigues J. Patterns of failure and survival for nonoperative treatment of stage c0 distal rectal cancer following neoadjuvant chemoradiation therapy. J Gastrointest Surg. 2006 Dec;10(10):1319-28; discussion 1328-9. doi: 10.1016/j.gassur.2006.09.005. PMID 17175450
- [Result] Habr-Gama A, Gama-Rodrigues J, Sao Juliao GP, Proscurshim I, Sabbagh C, Lynn PB, Perez RO. Local recurrence after complete clinical response and watch and wait in rectal cancer after neoadjuvant chemoradiation: impact of salvage therapy on local disease control. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):822-8. doi: 10.1016/j.ijrobp.2013.12.012. Epub 2014 Feb 1. PMID 24495589
- [Result] van der Valk MJM, Hilling DE, Bastiaannet E, Meershoek-Klein Kranenbarg E, Beets GL, Figueiredo NL, Habr-Gama A, Perez RO, Renehan AG, van de Velde CJH; IWWD Consortium. Long-term outcomes of clinical complete responders after neoadjuvant treatment for rectal cancer in the International Watch & Wait Database (IWWD): an international multicentre registry study. Lancet. 2018 Jun 23;391(10139):2537-2545. doi: 10.1016/S0140-6736(18)31078-X. PMID 29976470
- [Result] Smith JJ, Strombom P, Chow OS, Roxburgh CS, Lynn P, Eaton A, Widmar M, Ganesh K, Yaeger R, Cercek A, Weiser MR, Nash GM, Guillem JG, Temple LKF, Chalasani SB, Fuqua JL, Petkovska I, Wu AJ, Reyngold M, Vakiani E, Shia J, Segal NH, Smith JD, Crane C, Gollub MJ, Gonen M, Saltz LB, Garcia-Aguilar J, Paty PB. Assessment of a Watch-and-Wait Strategy for Rectal Cancer in Patients With a Complete Response After Neoadjuvant Therapy. JAMA Oncol. 2019 Apr 1;5(4):e185896. doi: 10.1001/jamaoncol.2018.5896. Epub 2019 Apr 11. PMID 30629084
- [Result] Appelt AL, Ploen J, Harling H, Jensen FS, Jensen LH, Jorgensen JC, Lindebjerg J, Rafaelsen SR, Jakobsen A. High-dose chemoradiotherapy and watchful waiting for distal rectal cancer: a prospective observational study. Lancet Oncol. 2015 Aug;16(8):919-27. doi: 10.1016/S1470-2045(15)00120-5. Epub 2015 Jul 5. PMID 26156652
- [Result] Dizdarevic E, Frostrup Hansen T, Ploen J, Henrik Jensen L, Lindebjerg J, Rafaelsen S, Jakobsen A, Appelt A. Long-Term Patient-Reported Outcomes After High-Dose Chemoradiation Therapy for Nonsurgical Management of Distal Rectal Cancer. Int J Radiat Oncol Biol Phys. 2020 Mar 1;106(3):556-563. doi: 10.1016/j.ijrobp.2019.10.046. Epub 2019 Nov 9. PMID 31707122
- [Result] Intven MPW, de Mol van Otterloo SR, Mook S, Doornaert PAH, de Groot-van Breugel EN, Sikkes GG, Willemsen-Bosman ME, van Zijp HM, Tijssen RHN. Online adaptive MR-guided radiotherapy for rectal cancer; feasibility of the workflow on a 1.5T MR-linac: clinical implementation and initial experience. Radiother Oncol. 2021 Jan;154:172-178. doi: 10.1016/j.radonc.2020.09.024. Epub 2020 Sep 22. PMID 32976875